CLINICAL TRIAL: NCT00202553
Title: Acceptability, Safety, Pharmacokinetics and Effects on Blood Pressure of a Daily Dose of 0.025 to 0.135 Milligram Per Kilogram of S90652, a Paediatric Formulation of Perindopril, in 2-16 Years Old Hypertensive Children - 3 Month Study
Brief Title: S90652 in Paediatric Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2-90652-001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Perindopril

INTERVENTIONS:
Drug: Perindopril

SUMMARY:
The aim of the study is to assess the acceptability, safety and pharmacokinetics and effects on blood pressure of a paediatric formulation of perindopril given in hypertensive children

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive children

Exclusion Criteria:

* Renal failure
* Unstable renal function
* Hyperkaliemia

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2003-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Safety assessed from the patient's (parents) complaints and the clinical follow-up

SECONDARY OUTCOMES:
Acceptability, efficacy, pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Niaudet, Pr, Study Chair — Hôpital Necker-Enfants Malades, Paris, France
Locations (1):
- Hôpital Necker Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies in patients:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com